CLINICAL TRIAL: NCT02393846
Title: Comparison of Topical Dexketoprofen Versus Placebo in Patients Presented With Ankle Sprain to the Emergency Department: A Randomised Placebo Controlled Trial
Brief Title: Topical Ketoprofen Versus Placebo in Patients With Ankle Sprain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Akdeniz University (Other)
Collaborators: Pamukkale University (Other)
Responsible Party: Principal Investigator, Cenker Eken, Associate Professor, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PAU2015/05
Record Dates: First submitted 2015-03-16; First posted 2015-03-20 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Ankle Sprain
Keywords: ankle sprain; topical ketoprofen; non-steroidal anti-inflammatory drug; emergency department
MeSH Terms: conditions — Ankle Injuries; Emergencies | interventions — ketoprofen topical gel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ketoprofen (Experimental): Topical ketoprofen (gel) is the experimental drug that is applied to the ankle in a dose of 2 gr.
  Interventions: Drug: Ketoprofen gel
- Placebo (Placebo Comparator): Topical placebo (gel) is identical in colour, form and smell with the ketoprofen gel.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketoprofen gel — Topical ketoprofen as used in gel form.
  Other Names: Fastjel
  Arms: ketoprofen
Drug: Placebo — Placebo gel which is identical in colour, form and smell compared to ketoprofen gel.
  Other Names: Placebo gel
  Arms: Placebo

SUMMARY:
The aim of this study is to analyse the effect of ketoprofen gel in patients presented with ankle sprain to the emergency department.

DETAILED DESCRIPTION:
Patients, 18-65 years old, presented with ankle sprain are enrolled into the study. Pain over 24 hours, pain intensity lower than 40 mm, allergy to the study drug, drug alcohol abuse and pregnancy or breastfeeding are the exclusion criteria. The study interventions are 2 gr of 2.5% ketoprofen gel versus placebo applied to the sprain area. The study drugs are identical in colour, form and smelling. After an eligible patient presented to the ED, the drug number from an opaque bag is determined by a nurse and then another nurse applies the study drug to the patient. Physicians, nurses and patients are blinded to the study drug. Pain intensity of patients is measured by visual analogue scale at baseline, 15th and 30th minutes after the administration.

ELIGIBILITY:
Inclusion Criteria:

* Patient presented with ankle sprain to the emergency department.
* Patients between 18-65 years old.

Exclusion Criteria:

* Pain over 24 hours,
* Pain intensity lower than 40 mm,
* allergy to the study drug,
* drug alcohol abuse
* pregnancy or breastfeeding are the exclusion criteria.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale | 30 minutes
  Pain intensity is measured by visual analogue scale at baseline, 15 and 30 minutes after the administration.

SECONDARY OUTCOMES:
Adverse effects | 30 minutes
  Adverse effects occurred during the study is recorded to the study form.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Serinken, MD, Study Chair — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)